CLINICAL TRIAL: NCT02925052
Title: Evaluation of the Gastric Tube Guide to Place Orogastric Tubes: : A Prospective, Randomized Trial
Brief Title: Evaluation of the Gastric Tube Guide to Place Orogastric Tubes
Acronym: GTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tim piepho, MD, PhD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTG-1
Record Dates: First submitted 2016-10-01; First posted 2016-10-05 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-03

CONDITIONS: Orogastric Tube Placement

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- GTG (Experimental): Gastric tube placement using the Gastric Tube Guide
  Interventions: Device: Gastric Tube Guide
- Conventional (Other): Gastric tube placement using a conventional method, according to local protocol.
  Interventions: Device: Conventional placement

INTERVENTIONS:
Device: Gastric Tube Guide
  Arms: GTG
Device: Conventional placement
  Arms: Conventional

SUMMARY:
A randomized controlled prospective study of orogastric tube placement with the Gastric Tube Guide vs conventional placement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* No concurrent participation in another study
* Capacity to consent
* Present written informed consent of the research participant
* Elective surgery in general anesthesia
* Required orogastric intubation

Exclusion Criteria:

* Existing pregnancy
* Emergency patients
* Preexisting pathological findings in the mouth, pharynx or esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Success | 180 seconds
  Overall Success after 180 seconds. Yes if a gastric tube was placed in time, no if not

SECONDARY OUTCOMES:
Attempts | 180 seconds
  Number of attempts that were necessary to place a gastric tube within 180 seconds
Time | 180 seconds
  Total time needed for gastric tube placement in seconds
Complications | 180 seconds
  Complications such as Bleeding, tooth damage, malposition (Scale yes or no)
Postoperative comfort | 24 hours
  Postoperative comfort is assessed using the postoperative section of the "core data set anaesthesia" from the German Society of Anaesthesiology and Intensive Care Medicine

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Mainz, Rhineland-Palatinate, Germany